CLINICAL TRIAL: NCT01451385
Title: An Open Label Safety Study of COV795 in Subjects With Osteoarthritis or Chronic Low Back Pain
Brief Title: Study of COV795 in Subjects With Osteoarthritis or Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COV15000181
Record Dates: First submitted 2011-09-29; First posted 2011-10-13 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis; Low Back Pain
MeSH Terms: conditions — Osteoarthritis; Low Back Pain | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- COV795 (Experimental): Participants receive 2 tablets of COV795 every 12 hours for up to 35 days
  Interventions: Drug: COV795

INTERVENTIONS:
Drug: COV795 — COV795 is a multilayer extended-release tablet for oral administration of oxycodone hydrochloride (15 mg) and acetaminophen (650 mg)
  Other Names: MNK795

SUMMARY:
The primary objective is to demonstrate the safety and tolerability of COV795 with up to 35 days use as evaluated by physical exam, vital signs, pulse oximetry, clinical laboratory tests, and other adverse events (AEs).

ELIGIBILITY:
Inclusion

1. Be considered in general good health based upon medical and surgical history, vital signs, pulse oximetry, physical exam, clinical lab tests, and electrocardiogram (ECG).
2. Be ≥18 years of age
3. Female subjects are eligible if not pregnant, not lactating or not planning to become pregnant within the next 2 months; surgically sterile or at least 2 years postmenopausal, or practicing an acceptable form of birth control for the duration of the study
4. Male subjects biologically capable of having children must agree to the use of a reliable method of birth control for the duration of the study
5. Have a clinical diagnosis of one of the following:

   * Osteoarthritis (OA) of the knee or hip for at least one year based on the American College of Rheumatology (ACR) criteria
   * Moderate to severe chronic lower back pain (CLBP), i.e. pain that occurs in an area with boundaries between the lowest rib and the crease of the buttocks that 1) must have been present for at least several hours a day for a minimum of 3 months, 2) is not due to a known malignancy, and 3) must be classified as non-neuropathic, neuropathic, or symptomatic for more than 6 months after lower back pain (LBP) surgery based on the Quebec Task Force Classification of Spinal Disorders
6. Have an average in-clinic pain score of ≥3 on the 11-point (0-10) numerical rating scale (NRS) as an average for the last 24 hours at screening visit.
7. Have a pain intensity score of ≥4 on NRS as an average for the last 24 hours at baseline visit.
8. Must, in the investigator's opinion, qualify for opioid therapy for their CLBP or OA.
9. Voluntarily provide written informed consent.

Exclusion

1. Have any clinically significant condition or unstable inter-current illness that would preclude study participation or interfere with the assessment of pain and other symptoms of CLBP or OA or would increase the risk of opioid-related AEs
2. Have an uncontrolled or poorly controlled major psychiatric condition, or have clinically significant anxiety or depression
3. Have an active malignancy or history of malignancy within 2 years
4. Have a history of seizures (except pediatric febrile seizures) or cognitive dysfunction
5. Have clinically significant ECG abnormalities or have uncontrolled hypo- or hypertension
6. Had arthroscopic or open surgery on either knee or hip selected as the primary OA study joint within 6 months
7. For CLBP, had a surgical procedure for back pain within 6 months
8. For CLBP participants, had a nerve or plexus block within 1 month or botulinum toxin injection in the lower back region within 3 months. For participants with OA of the selected primary joint, had joint injection within 1 month prior to Screening Visit 1.
9. Had surgical implants of either the knee or hip selected as the primary OA joint
10. Had gastric reduction surgery
11. Have been taking opioids in equivalents to more than 20 mg oxycodone hydrochloride (OC) or more than 40 mg morphine sulfate (MS) orally per day, or have been taking opioid medications 4 times a week or more
12. Unable to discontinue use of prohibited medications
13. Have a known allergy or hypersensitivity to opioids, OC, acetaminophen (APAP) or ibuprofen.
14. Have abnormal clinical laboratory tests at screening
15. Have a history of substance or alcohol abuse
16. Have positive screening labs for human immunodeficiency virus (HIV), Hepatitis B and/or Hepatitis C
17. Have a positive urine drug test for alcohol, illicit drugs, or controlled substances other than those prescribed medications
18. Have previously participated in a clinical trial using COV795
19. Received any investigational drugs or devices in the past 4 weeks
20. History of spinal stenosis
21. Other criteria as specified in the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2011-09-20; Primary Completion 2012-06-18 (Actual); Study Completion 2012-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Genova Clinical Research, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Research Institute, Anaheim, California
  - United Clinical Research Center, Inc., Anaheim, California
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - Catalina Research Institute, LLC, Chino, California
  - Synergy Escondido Clinical Research, Escondido, California
  - Convergys Clinical Research, Inc., Fresno, California
  - Triwest Research Associates, La Mesa, California
  - Skyline Research, Inc., Long Beach, California
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Avail Clinical Research, DeLand, Florida
  - Eastern Research, Hialeah, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Compass Research East, LLC, Oviedo, Florida
  - Gold Coast Research LLC, Plantation, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Sarasota Pain Medicine Research, LLC, Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Drug Studies America, Marietta, Georgia
  - Better Health Clinical Research, Newnan, Georgia
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - International Clinical Research Institute, Leawood, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - QUEST Research Institute, Bingham Farms, Michigan
  - Sundance Clinical Research, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Premier Research, Trenton, New Jersey
  - Peters Medical Research, High Point, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Hightop Medical Research Center/Hilltop Physicians Inc., Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Allegheny Pain Management, Altoona, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - Austin Diagnostic Clinic, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - Optimum Clinical Research, Inc., Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a screening period of up to 14 days, enrolled participants began treatment
Groups:
- All Participants: All participants receive 2 tablets of COV795 every 12 hours for up to 35 days
Period: Overall Study
Arm/Group | All Participants
Started | 376
Completed | 285
Not Completed | 91

BASELINE CHARACTERISTICS:
Population: All participants = safety population
Arm/Group | All Participants
Number analyzed (Participants) | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58
  Not Hispanic or Latino | 318
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 62
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 75
  White | 237
  More than one race | 0
  Unknown or Not Reported | 1
Modified Brief Pain Index - Short Form: Pain Intensity [Mean (Standard Deviation); unit: score on a scale] — Participants rate their pain on a scale from 0 = no pain to 10 = pain as bad as you can imagine
  score on a scale
    Worst pain in last 24 hours | 7.6 (1.32)
    Least pain in last 24 hours | 5.6 (1.94)
    Average pain in the last 24 hours | 6.7 (1.38)
    Pain right now | 6.7 (1.64)
Modified Brief Pain Inventory-Short Form: Percent Pain Relief from Medication [Mean (Standard Deviation); unit: percentage pain relief from medication] — Participants rate percent pain relief from medication on a scale from 0% (no relief) to 100% (complete relief)
  percentage pain relief from medication | 13.2 (21.93)
Modified Brief Pain Inventory-Short Form: Pain Interference Scores [Mean (Standard Deviation); unit: score on a scale] — Participants answer several questions about how much the pain interferes with their quality of life. The answers range from 0 = no interference to 10=completely interferes, and the average score for all the questions is recorded.
  score on a scale | 5.4 (2.03)
Western Ontario and McMaster U. Scores for Participants With Osteoarthritis (OA) of the Hip or Knee [Mean (Standard Deviation); unit: score on a scale] — Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC pain score ranges from 0 to 20, with higher scores representing worse pain. Population: Only participants with OA of the hip or knee were included in this outcome measure
  score on a scale
    number analyzed (Participants) | 140
    (all) | 11.74 (2.971)
WOMAC Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Stiffness Score [Mean (Standard Deviation); unit: score on a scale] — Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC stiffness score ranges from 0 to 8, with higher scores representing worse stiffness. Population: Participants in the safety population with OA of the hip or knee
  score on a scale
    number analyzed (Participants) | 140
    (all) | 4.94 (1.254)
WOMAC Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Physical Function [Mean (Standard Deviation); unit: score on a scale] — Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC physical function score ranges from 0 to 68, with higher scores representing worse functional limitations. Population: Participants in the safety population with OA of the hip or knee
  score on a scale
    number analyzed (Participants) | 140
    (all) | 38.96 (9.863)
WOMAC Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Total Score [Mean (Standard Deviation); unit: score on a scale] — Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC total score ranges from 0 to 96, with higher scores representing worse pain/disability. Population: Participants in the safety population with OA of the hip or knee
  score on a scale
    number analyzed (Participants) | 140
    (all) | 55.63 (13.251)
Roland-Morris Low Back Pain and Disability Scores for Participants with Chronic Low Back Pain [Mean (Standard Deviation); unit: score on a scale] — Roland-Morris Low Back Pain and Disability Scores for participants with chronic low back pain range from 0 to 24, with higher scores representing greater disability. Population: Participants in the safety population with chronic low back pain
  score on a scale
    number analyzed (Participants) | 235
    (all) | 10.9 (5.27)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Adverse Events (AEs)
Description: Collection of AEs began with subject's signing of the informed consent form, continued throughout the trial, and ended 7 days following the last dose of study drug, or at early termination. Treatment emergent AEs (TEAEs) are AEs that occurred after the first dose of study drug. TEAEs leading to discontinuation include 2 subjects who died (deaths not related to study drug). Clinically significant changes in values from physical exam, vital signs, clinical laboratory tests, and pulse oximetry were included as treatment emergent adverse events (TEAEs).
Time Frame: 5 Weeks
Population: All participants = safety population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 376
Participants
  Had any TEAE | 235
  Had a Severe TEAE | 17
  Had a TEAE related to study medication | 200
  Had a Serious AE | 4
  Died | 2
  Had a TEAE leading to discontinuation | 73

2. Secondary Outcome: Modified Brief Pain Index - Short Form: Pain Intensity
Description: Participants rate their pain on a score from 0=no pain to 10=pain as bad as you can imagine
Time Frame: at end of treatment (within 5 weeks)
Population: All participants = safety population with a score at end of treatment (week 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 359
score on a scale
  Worst pain in the last 24 hours | 4.0 (2.58)
  Least pain in last 24 hours | 2.4 (2.13)
  Average pain in the last 24 hours | 3.2 (2.25)
  Pain right now | 2.8 (2.36)

3. Secondary Outcome: Modified Brief Pain Index - Short Form: Percent Pain Relief From Medication
Description: Participants rate percent pain relief from medication on a scale from 0% (no relief) to 100% (complete relief)
Time Frame: at end of treatment (within 5 weeks)
Population: Safety population with a score at end of treatment
Measure: Mean (Standard Deviation); unit: percentage of relief from medication
Arm/Group | All Participants
Number analyzed (Participants) | 359
percentage of relief from medication | 67.7 (28.47)

4. Secondary Outcome: Modified Brief Pain Inventory-Short Form: Pain Interference Scores
Description: Participants answer several questions about how much the pain interferes with their quality of life. The answers range from 0 = no interference to 10=completely interferes, and the average score for all the questions is recorded.
Time Frame: at end of treatment (within 5 weeks)
Population: Safety population with a score at end of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 359
score on a scale | 2.2 (2.22)

5. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Pain Score
Description: Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC pain score ranges from 0 to 20, with higher scores representing worse pain.
Time Frame: End of treatment (within 5 weeks)
Population: Participants in the safety population with OA of the hip or knee and a score at end of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 134
score on a scale | 6.22 (4.016)

6. Secondary Outcome: WOMAC Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Stiffness Score
Description: Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC stiffness score ranges from 0 to 8, with higher scores representing worse stiffness.
Time Frame: End of treatment (within 5 weeks)
Population: Participants in the safety population with OA of the hip or knee and a score at end of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 134
score on a scale | 2.84 (1.713)

7. Secondary Outcome: WOMAC Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Physical Function Score
Description: Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC physical function score ranges from 0 to 68, with higher scores representing worse functional limitations.
Time Frame: End of treatment (within 5 weeks)
Population: Participants in the safety population with OA of the hip or knee and a score at end of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 134
score on a scale | 21.30 (13.180)

8. Secondary Outcome: WOMAC Questionnaire for Participants With Osteoarthritis (OA) of the Hip or Knee: Total Score
Description: Disease-specific quality of life is assessed using the WOMAC questionnaire (48-hour version) for participants with osteoarthritis (OA) of the hip or knee. The WOMAC total score ranges from 0 to 96, with higher scores representing worse pain/disability.
Time Frame: End of treatment (within 5 weeks)
Population: Participants in the safety population with OA of the hip or knee and a score at end of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 134
score on a scale | 30.35 (18.450)

9. Secondary Outcome: Roland-Morris Low Back Pain and Disability Scores for Participants With Chronic Low Back Pain
Description: Roland-Morris Low Back Pain and Disability Scores for participants with chronic low back pain range from 0 to 24, with higher scores representing greater disability.
Time Frame: End of treatment (within 5 weeks)
Population: Participants in the safety population with chronic low back pain and a score at end of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 224
score on a scale | 6.1 (5.75)

ADVERSE EVENTS:
Time Frame: From screening to follow-up, up to 45 days
Description: All treatment-emergent AEs are listed in the table of Other (Not Including Serious) Adverse Events
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 2/376
Serious Adverse Events (participants affected / at risk) | 4/376
Other Adverse Events (participants affected / at risk) | 235/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=376)
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=376)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Diplopia (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 42
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 6
Infrequent bowel movements (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 87
Oesophageal spasm (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 57
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Crepitations (General disorders) | 1
Fatigue (General disorders) | 8
Feeling jittery (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 1
Thirst (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Body tinea (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 5
Vaginal infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 5
Liver function test abnormal (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Fluid retention (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Balance disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 56
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 19
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 43
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 1
Cyclothymic disorder (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 2
Dysphoria (Psychiatric disorders) | 1
Euphoric mood (Psychiatric disorders) | 4
Hypervigilance (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 6
Middle insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 2
Withdrawal syndrome (Psychiatric disorders) | 1
Bladder discomfort (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Leukocyturia (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urine flow decreased (Renal and urinary disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 27
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 3
Hot flush (Vascular disorders) | 6
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes